CLINICAL TRIAL: NCT07262827
Title: A Pre-market, Prospective, Within-subject, Open-label, Interventional Investigation of Acceptance and Performance of Wireless Streaming Via Low Energy Audio Introduced Into the Firmware of the Nucleus 8 and Kanso 3 Sound Processors Worn by Experienced Adult Cochlear Implant Recipients
Brief Title: Investigating the Acceptance and Performance of Low Energy Audio Streaming in Nucleus 8 and Kanso 3 Sound Processors by Experienced Cochlear Implant Users
Acronym: STREAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLTD5844
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cochlear Implant Users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Experimental): Participants will be fit with either Nucleus 8 or Kanso 3 Sound Processors with LE Audio investigational firmware. Comparisons will be made within-participant with repeated measures for each of the speech perception scores in noise conditions.
  Interventions: Device: Nucleus 8 Sound Processor streaming via MultiMic+; Device: Nucleus 8 Sound Processor microphones; Device: Nucleus 8 Sound Processor streaming via Roger 20; Device: Kanso 3 Sound Processor streaming via Multi-Mic+; Device: Kanso 3 Sound Processor microphone

INTERVENTIONS:
Device: Nucleus 8 Sound Processor streaming via MultiMic+ — The Nucleus 8 Sound Processor streaming audio via the Multi-Mic+ wireless microphone accessory.
Device: Nucleus 8 Sound Processor microphones — Nucleus 8 Sound Processor streaming via the Nucleus 8 Sound Processor microphones (SCAN 2).
Device: Nucleus 8 Sound Processor streaming via Roger 20 — Nucleus 8 Sound Processor streaming audio via the Roger 20 wireless microphone accessory.
Device: Kanso 3 Sound Processor streaming via Multi-Mic+ — Kanso 3 Sound Processor streaming audio via the Multi-Mic+ wireless microphone accessory. This includes the Kanso 3 Nexa Sound Processor.
Device: Kanso 3 Sound Processor microphone — Kanso 3 Sound Processor streaming audio via the Kanso 3 Sound Processor microphones (SCAN 2). This includes the Kanso 3 Nexa Sound Processor.

SUMMARY:
This study aims to investigate acceptance and performance of the Bluetooth Low Energy Audio-enabled (LE Audio) firmware in the Nucleus 8 Processing Unit, Kanso 3 Nexa Sound Processor, and the Kanso 3 Sound Processor. The investigation includes actual use (take home) of LE Audio firmware releases and the new GN ReSound LE Audio wireless accessories, including the Multi-Mic+, for use in the real-world. Using the final versions of firmware, speech perception performance in noise will be investigated using the Nucleus 8 and Kanso 3 Sound Processors streaming via a Multi-Mic+.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Implanted with at least one of the CI1000 Series, CI600 Series, CI500 Series, Freedom Series or N24 Series cochlear hearing implants.
3. At least 3 months experience with a cochlear hearing implant
4. Demonstrated ability to score 30% or more at +15 SNR with Cochlear implant alone on a sentence in noise test.
5. Willingness to participate in and to comply with all requirements of the protocol
6. Fluent speaker in English as determined by the investigator
7. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Additional disabilities that would prevent participation in evaluations
2. Unrealistic expectations on the part of the participant, regarding the possible benefits, risks and limitations that are inherent to the procedures
3. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
5. Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by Investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Paired difference in City University of New York (CUNY) Sentences scores (% words correct) in classroom-like noise between the Nucleus 8 streaming via Multi-Mic+ and Nucleus 8 processor microphones (SCAN 2) at 0 dB SNR in 65 dB SPL | At ad-hoc visits between enrolment and 12 months

SECONDARY OUTCOMES:
Paired difference in CUNY Sentences scores (% words correct) in classroom-like noise between Nucleus 8 streaming via the Multi-Mic+ and Nucleus 8 streaming via the Roger 20 system at -15 dB SNR in 65 dB SPL | At ad-hoc visits between enrolment and 12 months
Paired difference in CUNY Sentences scores (% words correct) in classroom-like noise between Kanso 3 streaming via Multi-Mic+ and Kanso 3 processor microphones (SCAN 2) at 0 dB SNR in 65 dB SPL | At ad-hoc visits between enrolment and 12 months
Ratings based on the Device Use Questionnaire after a minimum of two weeks actual-use of the new GN ReSound accessories in the real-world environment | At ad-hoc visits between enrolment and 12 months
  The custom device use questionnaire is designed to collect information regarding the participants' experience using the research sound processors with the interventional accessories using a 5-point Likert scale (very satisfied, satisfied, neither dissatisfied nor satisfied, dissatisfied, very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Limited, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.